CLINICAL TRIAL: NCT00393536
Title: A Pragmatic Randomized Controlled Trial of Untargeted Educational Outreach Visiting Delivered by Pharmaceutical Advisers in Primary Care.
Brief Title: Study of Whether Educational Visits to Primary Care Professionals Improves the Quality of Care They Provide.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UEOVPAPHC-01
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: Depression
Keywords: Depression; Guidelines; Educational outreach visiting; Prescribing
MeSH Terms: conditions — Depression

INTERVENTIONS:
Behavioral: Educational outreach visiting

SUMMARY:
The purpose of this study is to find out whether educational visits by Pharmacists, who are already employed as advisers in health organisations, improve the prescribing habits of primary care doctors.

DETAILED DESCRIPTION:
Background There is increasing evidence that clinical guidelines can lead to improvements in both the process and outcome of care[1]. They figure prominently within the UK, particularly since the inception of the Scottish Intercollegiate Guidelines Network (SIGN) and the National Institute for Health and Clinical Excellence (NICE). However, clinical guidelines are not self-implementing and there is a growing body of research that demonstrates the effectiveness of various implementation strategies[1]. This has suggested that while the commonly used strategy of the postal distribution of educational materials alone may change clinician's behaviour it is unlikely to lead to large changes in practice. Educational outreach visits, using a trained person to meet face-to-face with a health care professional to provide information, may improve practice, especially prescribing behaviour[1,2]. Previous studies of the effectiveness of outreach visiting in the UK NHS have used local pharmacists as the visitors[3,4]. All Primary Care Trusts (PCTs) in England employ Pharmaceutical Advisers who are pharmacists whose role is to provide, from a wide clinical and health service management perspective, advice on prescribing and related areas to general practitioners (GPs). Pharmaceutical Advisers routinely visit general practices and are seen as change agents; however, the formal delivery of educational outreach by them has not been evaluated.

In 1996, the then Newcastle and North Tyneside Health Authority established a Clinical Effectiveness Unit. The remit of the Unit was to provide support to local health care teams in primary and secondary care, with the aim of promoting clinical effectiveness and encouraging the use of best evidence in daily practice through systematic, evidence-based approaches to guideline implementation. The strategy adopted by the Clinical Effectiveness Unit was to concentrate on five clinical areas. These were selected by a multi-disciplinary steering group using explicit criteria (evidence of inappropriate variation in practice; a good evidence base for what should be done; the clinical area should be a source of significant morbidity or mortality; large cost implications in the management of the topic). Depression was one of the clinical areas chosen.

The aim of this study was, for the choice of antidepressants for the management of depression, to evaluate, within a pragmatic cluster randomized controlled trial, the effectiveness of outreach visiting by existing Pharmaceutical Advisers in addition to the postal distribution of educational materials.

Methods Within a pragmatic randomized controlled trial, involving all general practices in two PCTs, routine methods were used to distribute guidelines for the choice of antidepressants for the management of depression. Intervention practices were offered two visits (most accepted only one) by their PCT Pharmaceutical Adviser who had been trained in the techniques of outreach visiting. The intervention was evaluated using level three Prescribing Analysis and Cost (PACT) data for antidepressant drugs for the six months during which the intervention was delivered and the subsequent 12 months

ELIGIBILITY:
Inclusion Criteria:

* all general practices in Newcastle and North Tyneside, England

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73
Dates: Start 1999-07; Study Completion 2000-12

PRIMARY OUTCOMES:
Usage of antidepressant drugs by type

SECONDARY OUTCOMES:
Costs of antidepressant drugs by type

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Eccles, MD, Principal Investigator — University of Newcastle Upon-Tyne
Locations (1):
- Institute of Health and Society, Newcastle upon Tyne, Tyne and Wear, United Kingdom